CLINICAL TRIAL: NCT02942225
Title: The Metabolome Profiling and Pathway Analysis of ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201601035RINA
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-03

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder; metabolomics; neuropsychological deficits; pathway analysis
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators will collect blood samples from each participant after 8-hour fasting. Blood samples will be transferred into evacuated tubes that contain anticoagulant sodium dihydrogen phosphate (EDTA), centrifuged at 2000g for 10 minutes at 4°C. Serum will be extracted and stored at -80°C for sample analysis. The collection of blood sample will be conducted at the NTUH.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ADHD group: Subjects with clinical diagnosis of ADHD according to the DSM-V criteria
- TD group: Typically development controls without lifetime diagnosis with ADHD

SUMMARY:
The purpose of this study is to understand the pathophysiological mechanisms of ADHD, especially the metabolomic pathway related to the behavioral/neuropsychological deficits of ADHD.

To identify specific metabolites that show significant differences between ADHD and control groups, both liquid chromatography-mass spectrometry and gas chromatography-mass spectrometry will be performed. In addition, the behavioral measures include ADHDRS-IV, SNAP-IV, CBCL, CGI-ADHD-S, SAICA, and Family APGAR-C. Neuropsychological testing, including CPT and CANTAB, will be performed. Conditional logistic regression and partial least squares discriminant analysis will be applied to identify significant metabolites for ADHD. Pathway enrichment and topology analyses will be conducted to evaluate the regulated pathways.

DETAILED DESCRIPTION:
Because attention deficit hyperactivity disorder (ADHD) is an early onset and long-term impairing disorder with tremendous impact on individuals, families, and societies, detection and diagnosis are very important for ADHD. Current diagnosis of ADHD relies mainly on clinical observation and interview tools that may involve a great subjective variability, and thus the investigation of objective biomarkers for ADHD is warranted. Metabolomics is the study of a biologic process involving all metabolites that are end products of the cellular process in a whole organism. Because metabolites represent the downstream expression of genome, transcriptome, and proteome, metabolomic profiles are more proximal to the behavioral phenotypes of ADHD. Analyzing metabolic differences between children with ADHD and healthy controls will provide insight into underlying disease pathology. To date, there has been no metabolomics study on ADHD. In this 3-year project, the investigators will perform a metabolomics analysis of serum to identify potential biomarkers for the behavioral and neuropsychological deficits of ADHD.

This is a 3-year project. After careful calculation of sample size, the investigators will recruit 120 drug-naïve children with ADHD, aged 7-18, and 120 healthy controls with matched age, sex and BMI. Using both liquid chromatography-mass spectrometry and gas chromatography-mass spectrometry, serum-based metabolomic profiling will be performed. The behavioral measures include ADHDRS-IV, SNAP-IV, CBCL, CGI-ADHD-S, SAICA, and Family APGAR-C. Neuropsychological testing, including CPT and CANTAB, will be performed. Conditional logistic regression and partial least squares discriminant analysis will be applied to identify significant metabolites for ADHD. Pathway enrichment and topology analyses will be conducted to evaluate the regulated pathways.

Using a matched study design, the investigators anticipate to identify specific metabolites that show significant differences between ADHD and control groups. In addition, results of pathway analysis may offer more biological understanding in explaining the underlying metabolic regulation among children with ADHD. This findings will significantly contribute to the knowledge of the pathophysiological mechanisms of ADHD, especially the metabolomic pathway related to the behavioral/neuropsychological deficits of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without any current or lifetime DSM-V psychiatric disorders based on the K-SADS-E interviews.

Exclusion Criteria:

* Participants who had any past or current medical or neurological illness, who currently took psychotropic medication, or whose intelligence quotient (IQ) score was less than 80 were excluded.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We plan to recruit 120 ADHD subjects and 120 control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Psychiatric interview | 1 hour
  Subjects will be interviewed by Chinese Version of the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E)

SECONDARY OUTCOMES:
Spatial working memory | 1.5 hours
  Subjects will be assessed by the Cambridge Neuropsychological Test Automated Battery (CANTAB)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yung Shang, MD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No